CLINICAL TRIAL: NCT02819414
Title: TIME TO RE-EVALUATE THE KINDER GENTLER APPROACH TO PATENT DUCTUS ARTERIOSUS (PDA) IN THE PRETERM NEONATE
Brief Title: Paracetamol Treatment of the Borderline Significant PDA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Cathy Hammerman, Director Div. Newborn Nurseries, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0174-16-SZMC
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): Treatment with placebo at a volume of 2.25 cc/kg/dose x 4/day to be given with feeds, or in place of feed when baby is receiving <2 cc/kg/feed.
  Interventions: Other: Placebo
- Treatment Group (Active Comparator): Treatment with paracetamol drops at 15 mg/kg/dose x 4/day. Drops will be diluted 1:15 in order to reduce osmolality. This will yield a dose of 2.25 ml/kg/dose, to be given with feeds, or in place of feed when baby is receiving <2 cc/kg/feed.
  Interventions: Drug: Paracetamol drops

INTERVENTIONS:
Drug: Paracetamol drops — 15 mg/kg/dose x 4/day diluted 1:15 yielding dose of 2.25 ml/kg/dose to be given for three days
  Other Names: Novimol
  Arms: Treatment Group
Other: Placebo — 2.25 ml/kg/dose x 4/day of sterile water to be given for three days
  Arms: Control Group

SUMMARY:
The therapeutic approach to the patent ductus arteriosus (PDA) in the premature neonate remains controversial. Currently it is generally accepted to treat only hemodynamically significant PDAs. The current investigation aims to study the effect of treatment on PDAs of borderline significance via a prospective, randomized controlled trial of paracetamol in this group.

DETAILED DESCRIPTION:
In the neonatal intensive care unit of the Shaare Zedek Medical Center, preterm babies <30 wks. GA, are studied echocardiographically on day of life 3-4. Pending parental informed consent, those diagnosed with a PDA of borderline significance will be randomized to receive either paracetamol or placebo for three days, followed by a repeat echocardiogram. If the PDA remains of borderline significance, the treatment will be continued for an additional 4 days (1 week total). Paracetamol levels and liver functions will be assessed after the third day. Babies will be followed until discharge for subsequent PDA pathology; respiratory distress and chronic lung disease [CLD]; necrotizing enterocolitis [NEC]; retinopathy of prematurity [ROP].

The investigators' primary goal is to demonstrate a decrease in the composite outcome of death or severe morbidity chronic lung disease [CLD], as shown by decreased time on supplemental oxygen and assisted ventilation.

Secondary goals:

* To demonstrate a decrease in subsequently diagnosed hs PDA, including

  * Decrease in the need for subsequent therapy for PDA closure
  * Decrease in surgical PDA ligations
* To demonstrate a decrease in necrotizing enterocolitis (NEC) and/or ROP with treatment.
* To demonstrate no adverse effect on blood flow in anterior cerebral, superior mesenteric and renal arteries.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates < 30 weeks' gestational age PDA of borderline significance

Exclusion Criteria:

* Infants not deemed likely to survive more than one week Infants with congenital heart malformations Infants with pulmonary hypertension and right to left ductal shunting

Ages: 3 Days to 6 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of death or severe morbidity chronic lung disease [CLD] | Day of life 3 until 40 weeks post-conception
  Chronic lung disease will be assessed by time on supplemental oxygen and assisted ventilation.

SECONDARY OUTCOMES:
Subsequently diagnosed hs PDA | Completion of study intervention until 40 weeks post-conception
  Will be assessed by subsequent need for medical or surgical intervention for closure of PDA
Subsequent incidence of necrotizing enterocolitis (NEC) and/or retinopathy of prematurity (ROP) | Completion of study intervention until 40 weeks post-conception
  Study infants will be followed clinically and any occurrence of NEC or ROP will be recorded with its level of significance (Bell staging for NEC and Stage of ROP)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Hammerman, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Terrin G, Conte F, Oncel MY, Scipione A, McNamara PJ, Simons S, Sinha R, Erdeve O, Tekgunduz KS, Dogan M, Kessel I, Hammerman C, Nadir E, Yurttutan S, Jasani B, Alan S, Manguso F, De Curtis M. Paracetamol for the treatment of patent ductus arteriosus in preterm neonates: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2016 Mar;101(2):F127-36. doi: 10.1136/archdischild-2014-307312. Epub 2015 Aug 17. PMID 26283668
- [Result] Hammerman C, Bin-Nun A, Markovitch E, Schimmel MS, Kaplan M, Fink D. Ductal closure with paracetamol: a surprising new approach to patent ductus arteriosus treatment. Pediatrics. 2011 Dec;128(6):e1618-21. doi: 10.1542/peds.2011-0359. Epub 2011 Nov 7. PMID 22065264